CLINICAL TRIAL: NCT04047719
Title: Pneumonia in the ImmunoCompromised - Use of the Karius Test for the Detection of Undiagnosed Pathogens
Acronym: PICKUP
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: KDC-010
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia, Bacterial; Pneumonia, Viral; Pneumonia Fungal; Pneumonia Cavitary; Immunocompromised Host
Keywords: Pneumonia; NGS; cell free DNA; microbial cell free DNA; immunocompromised
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia, Viral; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intent-to-Diagnose Population: All subjects enrolled in the study that have at least one Karius Test with a valid result
  Interventions: Diagnostic Test: Karius Test

INTERVENTIONS:
Diagnostic Test: Karius Test — Karius Test for detection of microbial cell free DNA (mcfDNA) in plasma

SUMMARY:
Given the need for a more sensitive pathogen detection test in patients with immunocompromised pneumonia, this study will evaluate the performance of the Karius Test, a novel NGS blood test for the diagnosis of infectious diseases. We will compare the performance of the Karius Test to the results of microbiologic tests obtained as part of usual care for immunocompromised patients undergoing evaluation for suspected pneumonia.

DETAILED DESCRIPTION:
Pneumonia is a major cause of morbidity and mortality in highly immunocompromised individuals such as patients with hematologic malignancies and/or hematopoietic stem cell transplant. These patients can be infected by a broad range of potential pathogens, including viral, bacterial, and fungal etiologies and sometimes with multiple pathogens simultaneously. Diagnostic testing often fails to identify a microbial etiology for lower respiratory illness even with bronchoalveolar lavage (BAL). In fact, culture methods, PCR, and antigen testing on BAL samples yields a positive result only 30-67% of the time. Additionally, Idiopathic Pulmonary Syndrome (IPS), a non-infectious pulmonary complication of transplant, can have many overlapping symptoms with infectious pneumonia. Treatment for IPS is administration of steroids which can exacerbate infections. Given these reasons, there is a need for better diagnostics to aid in the management of immunocompromised patients with pneumonia.

Karius has developed a microbial cell-free plasma next-generation sequencing test for pathogen detection capable of detecting >1,000 organisms including DNA viruses, bacteria, yeasts, molds, and other eukaryotic pathogens. The test is performed in a CLIA-certified/CAP-accredited laboratory with results typically provided within one day from sample receipt. Given the need for a more sensitive diagnostic test for pneumonia in this population, we are evaluating the performance of the Karius Test for pathogen detection.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the criteria in Section A and all of the criteria in either Section B, Section C or Section D.

Section A:

1. Patient is ≥ 18 years of age.
2. Is currently admitted to the hospital.
3. Has a suspected infectious pneumonia warranting diagnostic evaluation and treatment.
4. Has undergone a diagnostic bronchoscopy for the evaluation of microbiologic etiology of pneumonia within 1 day prior to or has a scheduled bronchoscopy within 5 days following enrollment.
5. Patient or patient's Legally Authorized Representative (LAR) has provided consent for the study.

Section B:

1. Has one of the following hematologic malignancies: Acute Lymphoblastic Leukemia (ALL), Acute Myelogenous Leukemia (AML), Myelodysplastic Syndrome (MDS), Lymphoma (any type), Multiple Myeloma (MM) or malignant transformation of Chronic Lymphocytic Leukemia (CLL/SLL).
2. Are immunocompromised defined as having at least one of the following:

   1. Received chemotherapy within the last 45 days.
   2. A relapse of hematologic malignancy for which chemotherapy treatment is anticipated within the next 45 days.
   3. ANC<500 for a minimum of 14 days and within 8 weeks prior to enrollment.

Section C:

1. Has undergone autologous hematopoietic stem cell transplantation (e.g. bone marrow transplantation) for one of the following hematologic malignancies: Acute Lymphoblastic Leukemia (ALL), Acute Myelogenous Leukemia (AML), Myelodysplastic Syndrome (MDS), Lymphoma (any type), or Multiple Myeloma (MM);), or malignant transformation of Chronic Lymphocytic Leukemia (CLL/SLL).
2. Are immunocompromised defined as having at least one of the following:

   1. Undergone autologous hematopoietic stem cell transplantation (HSCT) within the past 6 months.
   2. Received chemotherapy within the last 45 days.
   3. A relapse of hematologic malignancy for which chemotherapy treatment is anticipated within the next 45 days.

Section D:

1. Has undergone allogeneic hematopoietic stem cell transplantation (e.g., bone marrow transplantation) for any clinical indication.
2. Are immunocompromised defined as having at least one of the following:

   1. Has undergone hematopoietic stem cell transplantation (HCST) within the past 1 year.
   2. Has active graft versus host disease (GVHD) requiring immunosuppressive pharmacologic treatment.

Exclusion Criteria:

1. Patient is moribund and, in the opinion of the treating physician, is not expected to survive >24 hours beyond the time of potential study enrollment visit.
2. Microbiologic etiology of index pneumonia event has already been identified per local Standard of Care testing.
3. Patient was previously enrolled in this study.
4. Patient has any condition that, in the opinion of the treating physician, will prevent the patient from completing the study. (Note: a qualified patient may still enroll in the study if they decline to have exploratory research sample collected.)
5. Patient is positive for SARS-COV-2 by any molecular testing within the 14 days prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immunocompromised adult patients being evaluated for pneumonia who have undergone hematopoietic stem cell transplantation for any clinical indication or are receiving active chemotherapy for treatment of a hematologic malignancy.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Additive clinical diagnostic value | 7 days
  Percent of patients with ≥1 pathogen identified by the Karius Test collected at enrollment that is adjudicated as a probable cause of the subject's index pneumonia event with no pathogen identified as a probable cause of the subject's index pneumonia event from an adjudicated composite of all microbiologic test results performed per Standard of Care with results available within 7 days of study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bergin, MD, Principal Investigator — Duke University
Locations (10):
- United States (10):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Department of Medicine, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Tulane Section of Infectious Disease, New Orleans, Louisiana
  - Weill Cornell Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Norton ME, Baer RJ, Wapner RJ, Kuppermann M, Jelliffe-Pawlowski LL, Currier RJ. Cell-free DNA vs sequential screening for the detection of fetal chromosomal abnormalities. Am J Obstet Gynecol. 2016 Jun;214(6):727.e1-6. doi: 10.1016/j.ajog.2015.12.018. Epub 2015 Dec 18. PMID 26709085
- [Background] Alix-Panabieres C, Pantel K. Clinical Applications of Circulating Tumor Cells and Circulating Tumor DNA as Liquid Biopsy. Cancer Discov. 2016 May;6(5):479-91. doi: 10.1158/2159-8290.CD-15-1483. Epub 2016 Mar 11. PMID 26969689
- [Background] Evans SE, Ost DE. Pneumonia in the neutropenic cancer patient. Curr Opin Pulm Med. 2015 May;21(3):260-71. doi: 10.1097/MCP.0000000000000156. PMID 25784246
- [Background] Schuster MG, Cleveland AA, Dubberke ER, Kauffman CA, Avery RK, Husain S, Paterson DL, Silveira FP, Chiller TM, Benedict K, Murphy K, Pappas PG. Infections in Hematopoietic Cell Transplant Recipients: Results From the Organ Transplant Infection Project, a Multicenter, Prospective, Cohort Study. Open Forum Infect Dis. 2017 Mar 22;4(2):ofx050. doi: 10.1093/ofid/ofx050. eCollection 2017 Spring. PMID 28491889
- [Background] Chen CS, Boeckh M, Seidel K, Clark JG, Kansu E, Madtes DK, Wagner JL, Witherspoon RP, Anasetti C, Appelbaum FR, Bensinger WI, Deeg HJ, Martin PJ, Sanders JE, Storb R, Storek J, Wade J, Siadak M, Flowers ME, Sullivan KM. Incidence, risk factors, and mortality from pneumonia developing late after hematopoietic stem cell transplantation. Bone Marrow Transplant. 2003 Sep;32(5):515-22. doi: 10.1038/sj.bmt.1704162. PMID 12942099
- [Background] Harris B, Geyer AI. Diagnostic Evaluation of Pulmonary Abnormalities in Patients with Hematologic Malignancies and Hematopoietic Cell Transplantation. Clin Chest Med. 2017 Jun;38(2):317-331. doi: 10.1016/j.ccm.2016.12.008. PMID 28477642
- [Background] Hohenthal U, Itala M, Salonen J, Sipila J, Rantakokko-Jalava K, Meurman O, Nikoskelainen J, Vainionpaa R, Kotilainen P. Bronchoalveolar lavage in immunocompromised patients with haematological malignancy--value of new microbiological methods. Eur J Haematol. 2005 Mar;74(3):203-11. doi: 10.1111/j.1600-0609.2004.00373.x. PMID 15693789
- [Background] Blauwkamp TA, Thair S, Rosen MJ, Blair L, Lindner MS, Vilfan ID, Kawli T, Christians FC, Venkatasubrahmanyam S, Wall GD, Cheung A, Rogers ZN, Meshulam-Simon G, Huijse L, Balakrishnan S, Quinn JV, Hollemon D, Hong DK, Vaughn ML, Kertesz M, Bercovici S, Wilber JC, Yang S. Analytical and clinical validation of a microbial cell-free DNA sequencing test for infectious disease. Nat Microbiol. 2019 Apr;4(4):663-674. doi: 10.1038/s41564-018-0349-6. Epub 2019 Feb 11. PMID 30742071
- [Derived] Bergin SP, Chemaly RF, Dadwal SS, Hill JA, Lee YJ, Haidar G, Luk A, Drelick A, Chin-Hong PV, Benamu E, Khawaja F, Nanayakkara D, Papanicolaou GA, Small CB, Fung M, Barron MA, Davis T, McClain MT, Maziarz EK, Madut DB, Bedoya AD, Gilstrap DL, Todd JL, Barkauskas CE, Bigelow R, Leimberger JD, Tsalik EL, Wolf O, Mughar M, Hollemon D, Duttagupta R, Lupu DS, Bercovici S, Perkins BA, Blauwkamp TA, Fowler VG Jr, Holland TL. Plasma Microbial Cell-Free DNA Sequencing in Immunocompromised Patients With Pneumonia: A Prospective Observational Study. Clin Infect Dis. 2024 Mar 20;78(3):775-784. doi: 10.1093/cid/ciad599. PMID 37815489